CLINICAL TRIAL: NCT06986525
Title: A Prospective Split-Mouth Clinical Study Comparing Coronally Advanced Flap and Tunnel Techniques Combined With Platelet-Rich Fibrin in the Treatment of Multiple Gingival Recessions
Brief Title: Clinical Evaluation of Two Different Surgical Techniques With PRF in the Treatment of Multiple Gingival Recessions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Gizem Torumtay Cin, Assoc. Prof. Dr., Pamukkale University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: E-60116787-020-365617
Record Dates: First submitted 2025-05-09; First posted 2025-05-23 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-05

CONDITIONS: Gingival Recession
Keywords: gingival recessions; platelet rich fibrin; root coverage
MeSH Terms: conditions — Gingival Recession | interventions — Prolactin-Releasing Hormone

STUDY DESIGN:
Intervention Model Description: Split-mouth randomized design. Each participant receives both interventions, one per side of the mouth.
Masking Description: The clinical examiner who recorded the outcome measures was blinded to the type of surgical technique applied on each side.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAF + PRF (Experimental): This group will receive coronally advanced flap (CAF) surgery combined with platelet-rich fibrin (PRF) for the treatment of multiple gingival recessions.
  Interventions: Procedure: CAF with PRF
- Tunnel + PRF (Experimental): This group will receive tunnel surgical technique combined with platelet-rich fibrin (PRF) for the treatment of multiple gingival recessions.
  Interventions: Procedure: Tunnel with PRF

INTERVENTIONS:
Procedure: CAF with PRF — Coronally advanced flap technique will be performed to reposition the gingival margin coronally. Platelet-rich fibrin (PRF) membranes will be placed over the exposed root surfaces and stabilized with sutures.
  Arms: CAF + PRF
Procedure: Tunnel with PRF — A tunnel or subgingival pouch will be created using microsurgical instruments without vertical incisions. Platelet-rich fibrin (PRF) membranes will be inserted into the tunnel and the gingival tissue will be advanced coronally and sutured to cover the recession.
  Arms: Tunnel + PRF

SUMMARY:
This prospective clinical study aims to evaluate and compare the effectiveness of coronally advanced flap (CAF) and tunnel techniques, both combined with platelet-rich fibrin (PRF), in the treatment of multiple Miller Class I-II gingival recessions. Eleven participants with bilateral defects will be treated using a split-mouth design. Periodontal parameters will be assessed at baseline, 3 months, and 6 months.

DETAILED DESCRIPTION:
The objective of this prospective clinical trial is to compare two mucogingival surgical techniques-coronally advanced flap (CAF) and tunnel technique-used in combination with platelet-rich fibrin (PRF) for treating multiple Miller Class I-II gingival recessions. Eleven systemically healthy participants with bilateral gingival recessions will be enrolled. CAF+PRF will be applied on one side, and Tunnel+PRF on the contralateral side. Clinical parameters including plaque index, gingival index, bleeding on probing, probing depth, clinical attachment level, recession height and width, and keratinized tissue height will be recorded at baseline, 3 months, and 6 months. Root coverage outcomes and clinical attachment gain will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Systemically healthy individuals
* Presence of bilateral Miller Class I-II multiple gingival recessions
* Good oral hygiene and willingness to follow instructions
* Signed informed consent

Exclusion Criteria:

* Use of tobacco or smoking
* Pregnancy or lactation
* Presence of systemic diseases affecting periodontal health
* Use of medications that may affect healing (e.g., corticosteroids)
* Periodontal surgery in the same area within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Change in Recession Height (RH) | Baseline and 6 Months
  Recession height will be measured in millimeters from the cementoenamel junction to the gingival margin using a periodontal probe at baseline and 6 months postoperatively.

SECONDARY OUTCOMES:
Change in Clinical Attachment Level (CAL) | Baseline, 3 Months, and 6 Months
  Clinical attachment level will be measured in millimeters using a periodontal probe to assess periodontal healing at different time points.

CONTACTS AND LOCATIONS:
Overall Officials: Gizem TORUMTAY CİN, Assoc. Prof. Dr., Study Director — Pamukkale University Faculty of Dentistry, Department of Periodontology
Locations (1):
- Pamukkale University, Faculty of Dentistry, Periodontology, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This study does not plan to share individual participant data (IPD).